CLINICAL TRIAL: NCT02987491
Title: Exercise and Insulin Signaling in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 7605
Record Dates: First submitted 2016-11-21; First posted 2016-12-09 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Insulin Sensitivity; Obesity; Sedentary Lifestyle
Keywords: exercise
MeSH Terms: conditions — Insulin Resistance; Obesity; Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Metabolic Study Day (Experimental): Participants will perform a single bout of moderate intensity exercise on a cycle ergometer for 60 minutes.
  A total of 3 muscle biopsies will be collected throughout the study day. Insulin sensitivity will be measured using a hyperinsulinemic-euglycemic clamp with glucose tracers.
  Interventions: Behavioral: Exercise
- Resting Metabolic Study Day (No Intervention): Participants will rest quietly in bed for 60 minutes and resting energy metabolism will be measured with a ventilated hood.
  A total of 3 muscle biopsies will be collected throughout the study day. Insulin sensitivity will be measured using a hyperinsulinemic-euglycemic clamp with glucose tracers.

INTERVENTIONS:
Behavioral: Exercise — Participants will perform 2 metabolic study days of either resting or acute bout of cycling exercise in a randomized cross-over design.
  Arms: Exercise Metabolic Study Day

SUMMARY:
Obesity is associated with a decrease in skeletal muscle insulin sensitivity. Aerobic exercise can increase insulin sensitivity in the few hours following exercise, however the cellular mechanisms are not completely understood. The current project is to investigate mechanisms of exercise improvements to skeletal muscle insulin sensitivity.

DETAILED DESCRIPTION:
Study Overview: We are investigating the mechanisms by which exercise improves the response of skeletal muscle to insulin in lean and obese adults. Participants will complete 4 study visits consisting of: 1) screening visit, 2) maximal exercise test visit, and then a randomized order of 3) a resting metabolic study visit, and 4) an exercise metabolic study visit. Metabolic study visits for resting and exercise conditions will be identical, other than remaining sedentary or performing exercise. Skeletal muscle biopsy samples will be collected during resting, immediately post-exercise and during insulin stimulated conditions.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* Aged 18-45 years
* Normal weight (body mass index [BMI] 18-26 kg/m2) or obese (BMI 30-46 kg/m2)
* Sedentary (< 1 hour of planned physical activity per week for ≥ 6 months)
* Weight stable (< 2 kg change in body mass for ≥ 6 months)
* Non-smokers (no tobacco or nicotine use for ≥ 1 year)

Exclusion Criteria:

* Hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure > 90mmHg)
* Chronic health condition including diabetes, cardiovascular disease, treated hypertension, cancer, anemia, uncontrolled hyper- or hypothyroidism.
* Pregnant, nursing, irregular menses or post-menopausal (if female)
* Hyperglycemia (fasting glucose >126 mg/dl)
* Hypercholesterolemia (fasting LDL>140mg/dl)
* Hemoglobin < 13.0 g/dl (males), < 11.5 g/dl (females)
* Compromised renal function (outside 135-145 mmol/L sodium, 3.5-5.1 mmol/L potassium)
* Lidocaine allergy
* Medications including β-blockers, angiotensin converting enzyme inhibitors, insulin, thiazolidinediones, metformin, sulfonylureas, chronic non-steroidal anti-inflammatory use, anti-coagulant (e.g. warfarin), current antibiotics, opiates, monoamine oxidase inhibitors, benzodiazepines, or others that may impact the study outcomes
* Any physical limitation that prevents a participant from safely completing the exercise test
* Due to the risks associated with the current protocol, individuals with a diminished capacity to consent will be excluded. Similarly, due to the need for constant, accurate participant monitoring during metabolic study activities, participants will need to clearly understand verbal and written English. Participants who cannot clearly understand verbal and written English will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle insulin sensitivity | 2 hours following rest or exercise
  Skeletal muscle insulin sensitivity will be measured by hyperinsulinemic-euglycemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Robinson, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newsom SA, Stierwalt HD, Ehrlicher SE, Robinson MM. Substrate-Specific Respiration of Isolated Skeletal Muscle Mitochondria after 1 h of Moderate Cycling in Sedentary Adults. Med Sci Sports Exerc. 2021 Jul 1;53(7):1375-1384. doi: 10.1249/MSS.0000000000002615. PMID 34127633
- [Derived] Stierwalt HD, Ehrlicher SE, Robinson MM, Newsom SA. Skeletal Muscle ACSL Isoforms Relate to Measures of Fat Metabolism in Humans. Med Sci Sports Exerc. 2021 Mar 1;53(3):624-632. doi: 10.1249/MSS.0000000000002487. PMID 32796254

DOCUMENTS (1):
  • Informed Consent Form (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT02987491/ICF_000.pdf